CLINICAL TRIAL: NCT04576130
Title: A Danish Study to Assess the Efficacy of Implantable Cardioverter Defibrillator in Patients with Coronary Artery Disease Resuscitated from Ventricular Fibrillation Who Receive Complete Revascularization
Brief Title: A Danish ICD-study in Patients with Coronary Artery Disease Resuscitated from Ventricular Fibrillation
Acronym: DanICD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Reza Jabbari, Principal investigator, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-20007332
Record Dates: First submitted 2020-09-29; First posted 2020-10-06 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease; Acute Myocardial Infarction; Ventricular Fibrillation; Ventricular Tachycardia, Sustained; Out-Of-Hospital Cardiac Arrest
Keywords: Revascularization; Percutaneous coronary intervention; Implantable cardioverter defibrillator
MeSH Terms: conditions — Coronary Artery Disease; Ventricular Fibrillation; Tachycardia, Ventricular; Out-of-Hospital Cardiac Arrest | interventions — Defibrillators, Implantable

STUDY DESIGN:
Intervention Model Description: Randomized, parallel-group, open-label, superiority trial with two arms with 1:1 randomization through an internet-based randomization module.
Masking Description: Treatment cannot be blinded, we will use several endpoints that do not require an endpoint committee evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ICD-implantation (Experimental): Implantation of an ICD either during admission or within 4 weeks after discharge from index event.
  Interventions: Device: Implantable cardioverter defibrillator
- Standard care (No Intervention): Guideline directed medical therapy

INTERVENTIONS:
Device: Implantable cardioverter defibrillator — Implantation of an ICD for secondary prevention
  Other Names: ICD
  Arms: ICD-implantation

SUMMARY:
DanICD is a randomized, controlled study to with the aim to assess whether there is a benefit of ICD-implantation in patients with coronary artery disease (including acute myocardial infarction), who survive cardiac arrest due to ventricular fibrillation/sustained ventricular tachycardia and undergo revascularization and with an LVEF above 35%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CAD and cardiac arrest due to VF/VT, where angiogram is performed with complete revascularization (PCI, CABG or hybrid coronary revascularization) before ICD implantation. Unfavorable artery for PCI (i.e., excessive vessel tortuosity or chronic total occlusion) or high-risk invasive treatment is not mandatory in order to achive complete revascularization.
* Age ≥18 years
* LVEF >35% at the time of discharge. The most recent LVEF assessment on which the current medical treatment will be based at the time of entry into the study will be used as baseline LVEF.

Exclusion Criteria:

* Non-ischemic cause of cardiac arrest (i.e. ion channel diseases, non-ischemic cardiomyopathy)
* Previous CABG within the last 3 months before index hospitalization
* Life expectancy less than 1 year or severe neurologic outcome
* Unable or unwilling to give informed consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2032-10 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 5 years
  The clinical event committee will aim to attribute the cause of death to the underlying disease process rather than the immediate mechanism. Mortality will be classified as cardiovascular and non-cardiovascular.

SECONDARY OUTCOMES:
All cause mortality | 1 year
Sudden cardiovascular death | 1 year
  Cardiovascular death fulfilling the following criteria:
  * In witnessed cases a change in cardiovascular status with time until death being <1 hour.
  * In unwitnessed cases <24 hours since last seen alive and functioning normal.
Cardiovascular death | 1 year
  Mortality is considered as cardiovascular unless it is clearly attributable to another cause and thus includes:
  * Death due to proximate cardiac cause (e.g. myocardial infarction, cardiac tamponade, worsening heart failure).
  * Death caused by non-coronary vascular conditions such as neurological events, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular disease.
  * All procedure-related deaths, including those related to a complication of the ICD-procedure or treatment for a complication of the procedure.
  * All valve-related deaths including structural or non-structural valve dysfunction or other valve-related adverse events.
  * Death of unknown or cardiac cause.

OTHER OUTCOMES:
Device revision or replacement due to infection or malfunction | 1 year
  Explorative outcome
Appropriate shock from an ICD (successfully treated VT/VF) | 1 year
  Explorative outcome
Inappropriate shock from an ICD (shock on non-VT/VF) | 1 year
  Explorative outcome
Register-based all cause mortality | 10 years
Register-based sudden cardiovascular death | 5 years
Register-based sudden cardiovascular death | 10 years
Register-based cardiovascular death | 5 years
Register-based cardiovascular death | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Reza Jabbari, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided